CLINICAL TRIAL: NCT04911257
Title: Multi Center, Prospective Evaluation for Clinical and Radiographic Outcomes Utilizing Stryker Spine Cervical and Lumbar Interbody Systems: Observational Post Market Clinical Follow up Study
Brief Title: Interbody Systems: Post Market Clinical Follow-up Study
Status: Terminated | Type: Observational
Why Stopped: Sponsor terminated the study
Sponsor: K2M, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-017
Record Dates: First submitted 2021-05-17; First posted 2021-06-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Disc Disease
Keywords: Spondylolisthesis; Degenerative Scoliosis; Retrolisthesis.
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Degenerate Disc Disease: Subjects who will undergo spinal fusion surgery utilizing Stryker Interbody Systems.
  Interventions: Device: Cervical or Lumbar Spinal fusion

INTERVENTIONS:
Device: Cervical or Lumbar Spinal fusion — This is a prospective, multi-center study of subjects who will undergo spinal fusion surgery utilizing certain Stryker Interbody Systems.

SUMMARY:
This is a prospective, multi-center study of subjects who will undergo spinal fusion surgery utilizing Stryker Interbody Systems that require post market clinical follow up (PMCF).

The primary study hypothesis for each system is that the mean change in NDI (cervical) or ODI (lumbar) from baseline to Month 12 < -10, that is, the mean improvement exceeds 10 points. In supporting analysis, the same hypotheses will be tested for mean change from baseline to 24 months to demonstrate durability of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Must be planned to undergo spinal fusion surgery utilizing Stryker Interbody Systems for on label indications, which are listed below as inclusion criteria.
2. Diagnosed with degenerative disc disease (DDD).

   Please note for Lumbar devices:
   * Can also be diagnosed with up to Grade 1 Spondylolisthesis and/or Degenerative Scoliosis. (Chesapeake is not indicated for degenerative scoliosis)
   * Cascadia/Mojave/ Sahara/ Monterey AL can also be diagnosed with up to Grade 1 Retrolisthesis.

   Outside of USA, Tritanium is indicated for use in patients with diagnosis of Degenerative Spine Disorders, Spine Revision, Discal and Vertebral Instability; and there is no restriction to Spondylolisthesis Grade.
3. Willingness and ability to comply with the requirements of the protocol including follow up requirements.
4. Willing and able to sign a study specific informed consent form.
5. Skeletally mature (age at least 18 years) and:

   1. Have had six months of lumbar non operative therapy.
   2. Have had six weeks of cervical non operative treatment.
6. Will undergo interbody fusion at one or two contiguous levels (Chesapeake Cervical Ti is only indicated for use at one level) at:

   1. L2 L5 for Cascadia lateral hyperlordotic (>22°l).
   2. L2 S1 for all other lumbar interbody systems.
   3. C2 T1 for cervical interbody systems.
7. Self reports Oswestry Disability Index (ODI) score 30% (raw score of 15/50) for lumbar patients and Neck Disability Index (NDI) score 30% (raw score of 15/50) for cervical patients at pre operative visit.

Exclusion Criteria:

1. Any condition where the implants interfere with anatomical structures or precludes the benefit of spinal surgery.
2. For the Tritanium and Monterey AL systems: Any neuromuscular deficit which places an unsafe load on the device during the healing period.
3. For the Cascadia, Chesapeake, Mojave and Sahara systems: Metabolic disorders of calcified tissues.
4. Biological factors such as smoking or using nonsteroidal anti inflammatory agents/ anticoagulants.
5. Immunosuppressive disorders.
6. Grossly distorted anatomy. N/A for Tritanium TL, Tritanium Cervical and Monterey AL
7. Inadequate tissue coverage or open wounds.
8. Infection at index level(s) at the time of surgery.
9. Patients with known sensitivity to materials in the device.
10. Has a neuromuscular disorder or mental condition (including general neurological conditions, mental illness, senility, and drug/alcohol abuse) which would create an unacceptable risk of fixation failure or complications in postoperative care or willingness to restrict activities or follow medical advice.
11. Obesity.
12. Other medical or surgical condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors, congenital abnormalities, elevation of sedimentation rate unexplained by other diseases, elevation of white blood cell count (WBC) or marked left shift in the WBC differential count.
13. For the Tritanium and Monterey AL systems: Any abnormality which affects the normal process of bone remodeling including, but not limited to severe osteoporosis involving the spine, bone absorption, osteopenia, primary or metastatic tumors involving the spine or certain metabolic disorders affecting osteogenesis.

    Please note for Tritanium cervical this also includes rapid joint disease, bone absorption, osteopenia, osteomalacia, and/or osteoporosis.
14. For the Tritanium, Monterey AL, Chesapeake and Sahara systems: Prior fusion at the level to be treated (as indicated in the IFU).
15. Pregnancy, or if the patient intends to become pregnant during the course of the study.
16. Incarcerated at the time of study enrollment.
17. Current participation in an investigational study that may impact study outcomes.
18. Involved in current or pending litigation regarding a spine surgery.
19. Receiving worker's compensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will include patients that present with on-label conditions that will be surgically treated by participating investigators.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Mean Oswestry Disability Index Change | 12 Months
  Oswestry Disability Index (ODI) (lumbar) improvement from baseline to 12 months. Scale of Oswestry Disability Index from 0-50, 0 meaning no disability.
Mean Neck Disability Index Change | 12 Months
  Neck Disability Index (NDI) (cervical) improvement from baseline to 12 months. Scale of Neck Disability Index from 0-50, 0 meaning no disability.

SECONDARY OUTCOMES:
Mean Oswestry Disability Index Change | 24 Months
  Oswestry Disability Index (ODI) (lumbar) change from baseline to 24 months. Scale of Oswestry Disability Index from 0-50, 0 meaning no disability.
Mean Neck Disability Index Change | 24 months
  Neck Disability Index (NDI) (cervical) change from baseline to 24 months. Scale of Neck Disability Index from 0-50, 0 meaning no disability.
Safety Events | 24 months
  The following safety events will be collected through 24 months, including the following: (MedDRA will be used to define these events)
  * Serious adverse events
  * Device-related adverse events
  * Procedure-related adverse events
  * Operative site adverse events
  * Secondary spine surgeries (secondary interventions)
  * Adverse event that negatively impacts the primary endpoint
Fusion Status | 3, 6, 12 and 24 months
  Fusion will be derived from a logical analysis of three component factors: angular motion, translational motion, and bridging bone. Each treated level must be considered fused in order for the subject to be considered a radiographic success.
Angular Motion | 3, 6, 12 and 24 months
  Angular Motion will be measured from lateral flexion-extension radiographs. Angular motion, also known as rotation, is defined as the change in angle between the adjacent endplates of the motion segment. Angular Motion will be reported in units of degrees
Translational Motion | 3, 6, 12 and 24 months
  Translational Motion will be measured from lateral flexion-extension radiographs Translational motion is defined as the displacement of the posterior-inferior corner of the superior vertebra in a direction defined parallel to the superior endplate of the inferior vertebra. Translational Motion - Cervical will be reported in units of millimeters and percentage (%) of the anteroposterior (AP) length of the superior endplate of the inferior vertebra.
Bridging Bone | 3, 6, 12 and 24 months
  Interbody Bridging Bone will be graded in accordance with the following definitions:
  1. Absent: No evidence of continuous bridging bone from endplate to endplate.
  2. Present: Presence of continuous bridging bone from endplate to endplate.
Disc Height | PreOp, 2 and 6 weeks, 3, 6, 12 and 24 months
  Disc Height will be calculated from neutral lateral radiographs. Disc Height will be reported in units of millimeters and percentage (%) of the AP length of the superior endplate of the inferior vertebra. Average Disc Height
Device Migration | 6 weeks, 3, 6, 12 and 24 months
  Migration will be assessed relative to the Week 2 time point or earliest available post-operative visit. Migration will be measured in millimeters.
Subsidence | 6 weeks, 3, 6, 12 and 24 months
  Subsidence will be assessed relative to the Week 2 time point or earliest available post-operative visit, Subsidence will be measured in millimeters.
Adjacent Segment Degeneration | 2 and 6 weeks, 3, 6, 12 and 24 months
  Adjacent Segment Degeneration will be assessed at the adjacent levels using the Kellgren-Lawrence Osteoarthritis Grade.
Device and Supplemental Fixation Breakage | 2 and 6 weeks, 3, 6, 12 and 24 months
  Device and Supplemental Fixation Breakage will be assessed via all available x-ray images
Visual Analogue Scale Pain Severity | PreOp, 2 and 6 weeks, 3, 6, 12 and 24 months
  A Visual Analogue Scale patient questionnaire will be used to define the pain in the specific regions (cervical or lumbar) in the course of the study. 0 will be defined as "no pain" and 10 the Worst Possible Pain.
EQ-5D | PreOp, 2 and 6 weeks, 3, 6, 12 and 24 months
  The EQ-5D questionnaire is a standard generic patient questionnaire used to determine the health-related quality of life changes in the course of the study.
Prolo Scale | PreOp, 2 and 6 weeks, 3, 6, 12 and 24 months
  The Prolo Scale is a 10-point scale consisting of only two questions evaluating the functional and economic status of the patient in the course of this study.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Spine Institute of Louisiana Foundation, Inc., Shreveport, Louisiana
  - Cleveland Clinic, Cleveland, Ohio
  - The Spine Clinic of Oklahoma City, Oklahoma City, Oklahoma
  - Inova Neurosciences Research, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No